CLINICAL TRIAL: NCT04168749
Title: Efficacy and Safety of Introducing an Industrially Prepared Ready-to-use 3-Chamber Bag as Parenteral Nutrition Formulation for Premature Infants in Our NICU
Brief Title: Efficacy and Safety of Industrially Prepared 3 Chamber Bag Parenteral Nutrition for Premature Infant
Acronym: ESIP3CB
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Centre Hospitalier Universitaire de Tivoli (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CHUTivoli
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Weight Gain; Intravenous Nutrition Adverse Reaction; Premature
MeSH Terms: conditions — Weight Gain; Premature Birth | interventions — Parenteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- local compounding group: the first 100 preterm babies born as from January 1 2015 with a birth weight between 1250-2000g that received at least 10 days of TPN.
- Numeta G13 group: the first 100 preterm babies as from January 1 2017 with a birth weight between 1250-2000g that received at least 10 days of TPN
  Interventions: Combination Product: Numeta G13

INTERVENTIONS:
Combination Product: Numeta G13 — 10 days
  Other Names: parenteral nutrition for premature infant
  Groups: Numeta G13 group

SUMMARY:
This study was designed to evaluate whether industrially prepared standardizing total parenteral nutrition is at least non-inferior to compounded TPN and provides nutritional intakes according to the new guidelines and provides the expected weight gain in preterm babies with a birth weight between 1250 and 2000g admitted in our NICU between 2015 & 2018

DETAILED DESCRIPTION:
Parenteral nutrition (PN) is mandatory in the nursing of very low birth weight ((V)LBW)) babies during the first weeks of life. Numerous discussions exist about the indication of individually tailored or standardized PN formula. (V)LBW babies are known as fragile unstable babies with special requirements. Many neonatal intensive care units (NICU) prefer a tailored prescription for that kind of patients. Making a daily individual tailored prescription is often complex for numerous reasons: it is time consuming, it may be source of faults and incompatibility, it needs a senior neonatologist to review the prescription and has to arrive during daytime hours at the pharmacy. Tailored PN is often administrated with a delay, as one can only prescribe having reviewed the results of blood sampling. This delay can range from 6 to 12 hours. Numeta G13°/0E is a standardized, industrial, ready to use PN specifically designed to meet the nutritional requirements of preterm newborn infants for whom enteral nutrition is not possible or insufficient. New Espghan guidelines were published in 2018 recommending nutritional intake targets of 2.5g-3.5 amino acids per kg/day and 90-120 kcal/kg/day. Our NICU wants to evaluate their compliance to these new guidelines. Before November 2016, it was common practice in CHU Tivoli to feed the preterm baby with a compounded binary TPN solution and lipids were administered separately in Y-line. In November 2016, we switched to an all-in-one TPN with standardized composition (Numeta G13%E, Baxter) Numeta G13°/0E is stored at room temperature and is ready to be infused in a few minutes. Numeta G13%E is presented in the form of a three-chamber bag (3CB) or a two chamber bag (2CB). The activation of the lipid bag is optional, resulting in a solution containing glucose, electrolytes, amino acids and (optionally) lipids. Additions of water, electrolytes in the bag or on the side help to customize the bag to the specific needs of newborns that need intensive care.

ELIGIBILITY:
Inclusion Criteria:

* premature patients in the NICUs with a birth weight between 1250 and 2000g

Exclusion Criteria:

* death or parenteral duration less than 10 days

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: premature patients in the NICUs with a birth weight between 1250 and 2000g
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
weight gain in grams | 6 weeks
  grams

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève Malfilâtre, Principal Investigator — Centre Hospitalier Universitaire de Tivoli
Locations (1):
- Geneviève Malfilâtre, Soignies, Belgium

IPD SHARING:
Plan to Share IPD: No